CLINICAL TRIAL: NCT06362954
Title: The Effect of Spasticity Severity on Peripheral Muscle Oxygenation in Hemiparetic Stroke Patients
Brief Title: Muscle Oxygenation and Spasticity in Hemiparetic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Ankara Medipol University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Selcan Suicmez, Research Assistant, Ankara Medipol University
Other Study IDs: GaziU-FTR-SS-01
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Hemiparesis;Poststroke/CVA; Spasticity as Sequela of Stroke
Keywords: stroke; paresis; spasticity; near-infrared spectroscopy; lower extremity
MeSH Terms: conditions — Stroke; Paresis; Muscle Spasticity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- High-Level Spasticity Group: Hemiparetic stroke patients with spasticity levels greater than or equal 2 on the Modified Ashworth Scale.
- Low-Level Spasticity Group: Hemiparetic stroke patients with spasticity levels less than 2 on the Modified Ashworth Scale.
- Control Group: Healthy individuals were included in the control group.

SUMMARY:
Conditions such as hemiparesis, sensory and motor impairment, perceptual impairment, cognitive impairment, aphasia, and dysphagia may be observed after stroke. Motor impairment after stroke may occur due to damage to any part of the brain related to motor control. There is much clinical evidence that damage to different parts of the sensorimotor cortex in humans affects other aspects of motor function. Loss of strength, spasticity, limb apraxia, loss of voluntary movements, Babinski sign, and motor neglect are typical motor deficits following a cortical lesion (upper motor neuron lesion). Post-stroke spasticity can be seen in 19% to 92% of stroke survivors. Post-stroke hemiparesis is a significant cause of morbidity and disability, along with abnormal muscle tone. It has also been recognized that post-stroke hemiparesis may occur without spasticity. Spasticity influences muscle hemodynamic and oxidative metabolism, but its impact on the balance between oxygen delivery and utilization is not well understood.

This study study aims to investigate the effect of spasticity severity on peripheral muscle oxygenation in patients with hemiparetic stroke.

DETAILED DESCRIPTION:
Conditions such as hemiparesis, sensory and motor impairment, perceptual impairment, cognitive impairment, aphasia, and dysphagia may be observed after stroke. Motor impairment after stroke may occur due to damage to any part of the brain related to motor control. There is much clinical evidence that damage to different parts of the sensorimotor cortex in humans affects other aspects of motor function. Loss of strength, spasticity, limb apraxia, loss of voluntary movements, Babinski sign, and motor neglect are typical motor deficits following a cortical lesion (upper motor neuron lesion). Post-stroke spasticity can be seen in 19% to 92% of stroke survivors. Post-stroke hemiparesis is a significant cause of morbidity and disability, along with abnormal muscle tone. It has also been recognized that post-stroke hemiparesis may occur without spasticity. Spasticity influences muscle hemodynamic and oxidative metabolism, but its impact on the balance between oxygen delivery and utilization is not well understood.

Motor deficits seen in stroke patients and the conditions caused by them cause various limitations in the daily life of patients and affect their participation in daily life and quality of life. Decreased involvement in daily life negatively affects patients both socially and financially. Evaluating and identifying the disorders, taking preventive and developmental measures, and establishing treatment programs are necessary to increase participation. Therefore, objective and accurate assessment significantly affects the progress of the process.

Medical and surgical treatment and physiotherapy and rehabilitation approaches constitute the basis of treatment in stroke disease. The treatment of patients is carried out using a multidisciplinary approach involving many fields, such as medical and surgical treatment, physiotherapy, and rehabilitation practices. For this reason, it is seen that the financial burden, which cannot be covered by the insurance system from time to time, is relatively high. This burden is gradually increasing in direct proportion to the needs of the patients. For this reason, it is essential to develop practices and strategies for the patient's objective and most accurate evaluation, follow the clinical course, and create the most appropriate treatment program.

Although it is not among the routine evaluation methods, considering the studies conducted, "muscle oxygenation" should be considered in the evaluation phase in line with the possibilities.

ELIGIBILITY:
Stroke patients were included if they had a confirmed diagnosis (≥6 months post-stroke), were ≥18 years old, had hemiparesis with ankle plantar flexor spasticity, a Chedoke-McMaster Stroke Assessment score of 2-6 (leg/foot), a Modified Rankin Scale score of ≤4, and calf adipose tissue thickness <20 mm. Healthy controls were age- and gender-matched, ≥18 years old, with calf adipose tissue thickness <20 mm.

Exclusion criteria included severe uncontrolled hypertension, cardiovascular conditions limiting exercise, unrelated neurological or psychiatric disorders, and sensory impairments affecting the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty patients with chronic hemiparetic stroke and 10 healthy controls was conducted at Gazi University, Faculty of Health Sciences, Outpatient Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Gastrocnemius Muscle Oxygenation | Day 1
  Gastrocnemius muscle oxygenation will be evaluated with Near-Infrared Spectroscopy at rest, during and after the 6-Minute Walk Test (6MWT) and the Stair Climbing Test (SCT).
Spasticity | Day 1
  Plantar flexor muscle spasticity on the affected side will be evaluated with Modified Ashworth Scale

SECONDARY OUTCOMES:
Motor Function | Day 1
  Motor function of the affected limb was assessed using the leg and foot sections of the Chedoke-McMaster Stroke Assessment (1-7 scale).
Disability Level | Day 1
  Disability level was determined using the Modified Rankin Scale, which ranges from 0 (no symptoms) to 6 (death).
6-Minute Walk Test | Day 1
  Submaximal functional capacity will be evaluated with 6-Minute Walk Test during muscle oxygenation measurement.
Stair Climbing Test | Day 1
  Maximal functional capacity will be evaluated with Stair Climbing Test during muscle oxygenation measurement.
Adipose tissue thickness | Day 1
  The skinfold thickness of gastrocnemius muscle was evaluated with a Skinfold Caliper. Adipose tissue thickness was obtained by dividing the skinfold thickness by two.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Faculty of Health, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suicmez S, Yazici G, Altiparmak T, Cagatay C, Batur-Caglayan HZ, Nazliel B. The effect of spasticity severity on peripheral muscle oxygenation in hemiparetic stroke patients: a cross-sectional study. Top Stroke Rehabil. 2026 Mar;33(2):164-174. doi: 10.1080/10749357.2025.2538520. Epub 2025 Jul 28. PMID 40717605